CLINICAL TRIAL: NCT01818245
Title: Effect of Injection Site on the Pharmacokinetics and Pharmacodynamics of Single Subcutaneous Doses of LY2605541 in Healthy Subjects, and Impact of Body Mass Index and Age on the Pharmacokinetics of LY2605541
Brief Title: A Study of LY2605541 in Healthy Participants and in the Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 12152; I2R-MC-BIDF (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY2605541

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2605541: Cohort A (Injection site: Abdomen) (Experimental): Participants ≤55 years of age will receive 1 subcutaneous (SC) injection of 0.5 Units per kilogram (U/kg) of LY2605541 in the abdominal wall on Day 1 in 1 of 3 treatment periods. There was a washout period of 16-28 days between each treatment period.
  Interventions: Drug: LY2605541
- LY2605541: Cohort A (Injection site: Upper Arm) (Experimental): Participants ≤55 years of age will receive 1 SC injection of 0.5 U/kg of LY2605541 in the upper arm on Day 1 in 1 of 3 treatment periods. There was a washout period of 16-28 days between each treatment period.
  Interventions: Drug: LY2605541
- LY2605541: Cohort A (Injection site: Thigh) (Experimental): Participants ≤55 years of age will receive 1 SC injection of 0.5 U/kg of LY2605541 in the thigh on Day 1 in 1 of 3 treatment periods. There was a washout period of 16-28 days between each treatment period.
  Interventions: Drug: LY2605541
- LY2605541: Cohort B (Injection site: Abdomen) (Experimental): Participants ≥65 years of age will receive 1 SC injection of 0.5 U/kg of LY2605541 in the abdominal wall on Day 1.
  Interventions: Drug: LY2605541

INTERVENTIONS:
Drug: LY2605541

SUMMARY:
This study will include 2 groups (cohorts) of participants:

In Cohort A, this study will look at the amount of LY2605541 that is present in the body after it is injected in 3 different locations in the body of the same participant. At least 16 days will pass between each injection.

In Cohort B, the study will look at how the body absorbs, distributes, and disposes of LY2605541 in participants aged 65 and over.

Participants may enroll in only one cohort.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: are overtly healthy male or female participants, as determined by medical history and physical examination, aged ≥18 to ≤55 years of age
* Cohort B: are male or female elderly (≥65 years of age) participants that are overtly healthy, or have stable, chronic medical conditions (including Type 2 Diabetes Mellitus [T2DM]) that, in the investigator's opinion, will not significantly alter the disposition of the drug, will not place the participant at increased risk by participating in the study, and will not interfere with interpretation of the data
* Male participants agree to use a reliable method of birth control during the study and for 3 months following the last dose of the investigational product
* Female participants are women of child-bearing potential who test negative for pregnancy at the time of screening based on a urine pregnancy test and agree to use a reliable method of birth control during the study and for 1 month following the last dose of the investigational product
* Female participants are post-menopausal women, or women not of child-bearing potential due to surgical sterilization (at least 3 months after surgical hysterectomy, or at least 3 months after bilateral oophorectomy or bilateral tubal ligation/occlusion with or without hysterectomy) confirmed by medical history, or menopause
* Have a body mass index (BMI) of 18.5 to 40 kilogram per meter square (kg/m^2), inclusive, at time of admission for Period 1
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are participants that intend to start a change in diet or lose weight during the study; participants will be expected to maintain their approximate current weight throughout the study
* Are excessive smokers (>10 cigarettes per day); participants who smoke ≤10 cigarettes per day must be able to stop smoking while residing at the clinical research unit (CRU)

Healthy Participants - Cohort A

* Have Type 1 Diabetes Mellitus (T1DM), Type 2 Diabetes Mellitus (T2DM), or a fasting blood glucose (BG) >110 milligrams per deciliter (mg/dL) (6.1 millimoles per liter [mmol/L]) with a glycated hemoglobin (HbA1c) of >6.2%
* Intend to use over-the-counter medication within the 7 days or prescription medication within 14 days prior to dosing (apart from contraceptive medication, vitamin/mineral supplements, occasional paracetamol, thyroxine replacement therapy, and hormone replacement therapy). Antihypertensive and lipid lowering agents are permitted, but must have been administered at stable dose(s) for at least 1 month.

Elderly Participants - Cohort B

* Have T1DM
* Are T2DM participants that require insulin treatment, or have a HbA1c of >10%
* Have started new chronic medication(s) or changed the dose of an existing chronic medication <1 month prior to dosing. Participants are permitted to continue ongoing chronic medications (for example antihypertensive agents, aspirin, non-steroidal anti-inflammatory drugs, lipid lowering agents, thyroxine, hormone replacement therapy, and/or oral anti-diabetic if participants have T2DM). Other stable chronic conditions may be permitted if deemed acceptable by the investigators and Lilly clinical pharmacologist or clinical research physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2605541: Cohort A (Participants ≤55 Years of Age): Participants ≤55 years of age were randomized to 1 of 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, or CBA), each of which was comprised of the same 3 interventions (A, B, and C). Each intervention was separated by a 16-28 day washout.
  Intervention A: participants ≤55 years of age received 1 subcutaneous (SC) injection of 0.5 Units per kilogram (U/kg) of LY2605541 in the abdominal wall on Day 1 of the treatment period.
  Intervention B: participants ≤55 years of age received 1 SC injection of 0.5 U/kg of LY2605541 in the upper arm on Day 1 of the treatment period.
  Intervention C: participants ≤55 years of age received 1 SC injection of 0.5 U/kg of LY2605541 in the thigh on Day 1 of the treatment period.
- LY2605541: Cohort B (Participants ≥65 Years of Age): Participants ≥65 years of age received 1 SC injection of 0.5 U/kg of LY2605541 in the abdominal wall on Day 1.
Period: Intervention A
Arm/Group | LY2605541: Cohort A (Participants ≤55 Years of Age) | LY2605541: Cohort B (Participants ≥65 Years of Age)
Started | 30 | 22 (Participants didn't participate in separate interventions and received 1 dose of LY2605541 on Day 1.)
Received One Dose of Study Drug | 30 | 22
Completed | 30 | 22
Not Completed | 0 | 0
Period: Washout (16-28 Days)
Arm/Group | LY2605541: Cohort A (Participants ≤55 Years of Age) | LY2605541: Cohort B (Participants ≥65 Years of Age)
Started | 30 | 0
Completed | 30 | 0
Not Completed | 0 | 0
Period: Intervention B
Arm/Group | LY2605541: Cohort A (Participants ≤55 Years of Age) | LY2605541: Cohort B (Participants ≥65 Years of Age)
Started | 30 | 0
Completed | 30 | 0
Not Completed | 0 | 0
Period: Washout (16-28 Days)
Arm/Group | LY2605541: Cohort A (Participants ≤55 Years of Age) | LY2605541: Cohort B (Participants ≥65 Years of Age)
Started | 30 | 0
Completed | 30 | 0
Not Completed | 0 | 0
Period: Intervention C
Arm/Group | LY2605541: Cohort A (Participants ≤55 Years of Age) | LY2605541: Cohort B (Participants ≥65 Years of Age)
Started | 30 | 0
Completed | 30 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY2605541: Cohort A (Participants ≤55 Years of Age): Participants ≤55 years of age were randomized to 1 of 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, or CBA), each of which was comprised of the same 3 interventions (A, B, and C). Each intervention was separated by a 16-28 day washout.
  Intervention A: participants ≤55 years of age received 1 SC injection of 0.5 U/kg of LY2605541 in the abdominal wall on Day 1 of the treatment period.
  Intervention B: participants ≤55 years of age received 1 SC injection of 0.5 U/kg of LY2605541 in the upper arm on Day 1 of the treatment period.
  Intervention C: participants ≤55 years of age received 1 SC injection of 0.5 U/kg of LY2605541 in the thigh on Day 1 of the treatment period.
- Total: Total of all reporting groups
Arm/Group | LY2605541: Cohort A (Participants ≤55 Years of Age) | LY2605541: Cohort B (Participants ≥65 Years of Age) | Total
Number analyzed (Participants) | 30 | 22 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (9.1) | 71.4 (6.3) | 51.7 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 20 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 26 | 21 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 7 | 23
  White | 10 | 15 | 25
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 22 | 52

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC): Injection Site (Arm and Thigh) Versus Abdominal Wall Injection (Cohort A)
Description: AUC from time zero to infinity (AUC(0-∞)) of LY2605541 was evaluated across injection sites (abdominal wall, arm, and thigh).
Time Frame: Predose and 2, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours postdose
Population: Participants in Cohort A who received LY2605541 and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles*hours/liter (pmol*h/L)
Groups:
- LY2605541: Cohort A (Injection Site: Abdomen): Participants ≤55 years of age will receive 1 SC injection of 0.5 U/kg of LY2605541 in the abdominal wall on Day 1 in 1 of 3 treatment periods.
- LY2605541: Cohort A (Injection Site: Upper Arm): Participants ≤55 years of age will receive 1 SC injection of 0.5 U/kg of LY2605541 in the upper arm on Day 1 in 1 of 3 treatment periods.
- LY2605541: Cohort A (Injection Site: Thigh): Participants ≤55 years of age will receive 1 SC injection of 0.5 U/kg of LY2605541 in the thigh on Day 1 in 1 of 3 treatment periods.
Arm/Group | LY2605541: Cohort A (Injection Site: Abdomen) | LY2605541: Cohort A (Injection Site: Upper Arm) | LY2605541: Cohort A (Injection Site: Thigh)
Number analyzed (Participants) | 30 | 30 | 30
picomoles*hours/liter (pmol*h/L) | 124000 (37) | 133000 (39) | 135000 (36)

2. Primary Outcome: Pharmacokinetics: Observed Maximum Plasma Concentration (Cmax): Injection Site (Arm and Thigh) Versus Abdominal Wall Injection (Cohort A)
Description: Cmax of LY2605541 was evaluated across injection sites (abdominal wall, arm, and thigh).
Time Frame: Predose and 2, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours postdose
Population: Participants in Cohort A who received LY2605541 and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles/liter (pmol/L)
Arm/Group | LY2605541: Cohort A (Injection Site: Abdomen) | LY2605541: Cohort A (Injection Site: Upper Arm) | LY2605541: Cohort A (Injection Site: Thigh)
Number analyzed (Participants) | 30 | 30 | 30
picomoles/liter (pmol/L) | 1839.17 (59) | 1700.68 (54) | 2027.99 (66)

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC): Elderly Participants (≥65 Years of Age) Versus Participants ≤55 Years of Age (Abdominal Injection)
Description: AUC(0-∞) for LY2605541 was evaluated.
Time Frame: Predose and 2, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours postdose
Population: Participants in Cohort A and B who received LY2605541 in the abdomen and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Arm/Group | LY2605541: Cohort A (Injection Site: Abdomen) | LY2605541: Cohort B (Injection Site: Abdomen)
Number analyzed (Participants) | 30 | 22
pmol*h/L | 124000 (37) | 134000 (30)

4. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax): Elderly Participants (≥65 Years of Age) Versus Participants ≤55 Years of Age (Abdominal Injection)
Description: Cmax of LY2605541 was evaluated.
Time Frame: Predose and 2, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours postdose
Population: Participants in Cohort A and B who received LY2605541 in the abdomen and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | LY2605541: Cohort A (Injection Site: Abdomen) | LY2605541: Cohort B (Injection Site: Abdomen)
Number analyzed (Participants) | 30 | 22
pmol/L | 1839.17 (59) | 1829.92 (49)

5. Secondary Outcome: Pharmacodynamics: Total Amount of Glucose Infused (Gtot): Injection Site (Arm and Thigh) Versus Abdominal Wall Injection (Cohort A)
Description: Gtot was evaluated across injection sites (abdominal wall, arm, and thigh).
Time Frame: Predose up to 24 hours post clamp procedure in all treatment periods
Population: Participants in Cohort A who received LY2605541 and had evaluable Gtot data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilograms (mg/kg)
Groups:
- LY2605541 - Cohort A (Injection Site: Abdomen): Participants ≤55 years of age will receive 1 SC injection of 0.5 U/kg of LY2605541 in the abdominal wall on Day 1 in 1 of 3 treatment periods.
Arm/Group | LY2605541 - Cohort A (Injection Site: Abdomen) | LY2605541: Cohort A (Injection Site: Upper Arm) | LY2605541: Cohort A (Injection Site: Thigh)
Number analyzed (Participants) | 29 | 30 | 29
milligrams/kilograms (mg/kg) | 674 (109) | 633 (102) | 454 (204)

6. Secondary Outcome: Pharmacodynamics: Maximum Glucose Infusion Rate (Rmax): Injection Site (Arm and Thigh) Versus Abdominal Wall Injection (Cohort A)
Description: Rmax was evaluated across injection sites (abdominal wall, arm, and thigh).
Time Frame: Predose up to 24 hours post clamp procedure in all treatment periods
Population: Participants in Cohort A who received LY2605541 and had evaluable Rmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/minute/kilogram (mg/min/kg)
Arm/Group | LY2605541: Cohort A (Injection Site: Abdomen) | LY2605541: Cohort A (Injection Site: Upper Arm) | LY2605541: Cohort A (Injection Site: Thigh)
Number analyzed (Participants) | 29 | 30 | 29
milligrams/minute/kilogram (mg/min/kg) | 0.944 (88) | 0.935 (83) | 0.738 (144)

ADVERSE EVENTS:
Arm/Group | LY2605541: Cohort A (Injection Site: Abdomen) | LY2605541: Cohort A (Injection Site: Upper Arm) | LY2605541: Cohort A (Injection Site: Thigh) | LY2605541: Cohort B (Injection Site: Abdomen)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/22
Other Adverse Events (participants affected / at risk) | 3/30 | 5/30 | 13/30 | 7/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541: Cohort A (Injection Site: Abdomen) (N=30) | LY2605541: Cohort A (Injection Site: Upper Arm) (N=30) | LY2605541: Cohort A (Injection Site: Thigh) (N=30) | LY2605541: Cohort B (Injection Site: Abdomen) (N=22)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 6 (7) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days